CLINICAL TRIAL: NCT01933776
Title: Clinical Safety Study of the Tdap Combined Vaccine (ADACEL™) as a Booster Dose in Healthy Adults and Children in China
Brief Title: Study of the Tdap Combined Vaccine (ADACEL™) as a Booster Dose in Healthy Adults and Children in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Td527; U1111-1127-7738 (Other: WHO)
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: Diphtheria; Tetanus; Pertussis; ADACEL®; Tdap vaccine
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Tetanus Toxoid; adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Adults (Experimental): Participants 18 through 64 years of age will receive a single booster dose of Tdap vaccine (ADACEL).
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Tdap
- Group 2: Children (Experimental): Participants 4 through 8 years of age will receive a single booster dose of Tdap vaccine (ADACEL)
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Tdap

INTERVENTIONS:
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Tdap — 0.5 mL, Intramuscular (IM)
  Other Names: ADACEL™
  Arms: Group 1: Adults
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Tdap — 0.5 mL, Intramuscular (IM)
  Other Names: ADACEL™
  Arms: Group 2: Children

SUMMARY:
The aim of the study is to assess the safety profile of ADACEL vaccine in a small number of participants in China.

Primary objective:

* To describe the safety in terms of occurrence of serious adverse reactions and grade 3 adverse reactions after administration of Sanofi Pasteur's Tdap vaccine (ADACEL) given as a single dose in 20 adults and 20 children.

Secondary objective:

* To describe the full reactogenicity profile after administration of sanofi pasteur's Tdap vaccine (ADACEL) given as a single dose in 20 adults and 20 children.

DETAILED DESCRIPTION:
Participants will be enrolled sequentially into the study groups to receive one dose of ADACEL at Day 0 (Visit 1) and will be followed-up for 28-35 days.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Aged 18 through 64 years on the day of inclusion Group 2: Aged 4 through 8 years on the day of inclusion
* Informed consent form signed by the subject (Group 1) or by the parent(s) or legal representative (Group 2)
* Subject (Group 1 and 2) and parent/legal representative (Group 2 only) able to attend all scheduled visits and to comply with all trial procedures
* Group 1 only: For a woman of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) from at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination
* Group 2 only: Written documentation of complete primary series and fourth dose of Diphtheria, Tetanus, Pertussis (DTP) vaccine as per China National Immunization Recommendations

Exclusion Criteria:

* Group 1 only: For a woman of child-bearing potential, known pregnancy or positive serum or urine pregnancy test
* Group 1 only: Currently breast-feeding a child
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine or to a vaccine containing any of the same substances
* Chronic illness that, in the opinion of the Investigator, is at a stage that could interfere with trial conduct or completion
* Group 1 only: Current alcohol abuse or drug addiction that may interfere with the ability to comply with trial procedures
* Receipt or planned receipt of any vaccine in the 4 weeks preceding or following trial vaccination, except for influenza vaccination, which may be received at least two weeks before the study vaccine
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C
* History of diphtheria, tetanus, or pertussis infection (confirmed either clinically, serologically or microbiologically)
* Previous fifth vaccination against pertussis disease and/or previous sixth vaccination against diphtheria and tetanus disease with either the trial vaccine or another vaccine (except Tetanus-prone wound management in Group 1)
* Subject at high risk for diphtheria, tetanus, or pertussis infection during the trial, including persons who have exposure (e.g., member of a household with another infected member, travelers to or residents of areas where one of this disease is hyperendemic or epidemic, or microbiologists routinely working with one of these pathogens,)
* Self-reported thrombocytopenia, bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Group 1 only: Subjects deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* History of contra-indication to vaccination with pertussis containing vaccine, including:
* Encephalopathy (eg, coma, decreased level of consciousness, prolonged seizures) within 7 days of a previous dose of a pertussis containing vaccine that is not attributable to another identifiable cause
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as immediate family members (i.e. husband, wife and their children, adopted or natural) of the employees or the Investigator.

Ages: 4 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Jiangsu, Jiangsu, China

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 27 August 2013 through 08 October 2013 at 1 clinic center in China.
Pre-assignment Details: A total of 40 participants who met all of the inclusion and none of the exclusion criteria were enrolled and vaccinated in this study.
Groups:
- ADACEL™ Vaccine Group 1 (Adults): Adults 18 through 64 years of age received a single booster dose of Tdap vaccine (ADACEL™)
- ADACEL™ Vaccine Group 2 (Children): Children 4 through 8 years of age received a single booster dose of Tdap vaccine (ADACEL™)
Period: Overall Study
Arm/Group | ADACEL™ Vaccine Group 1 (Adults) | ADACEL™ Vaccine Group 2 (Children)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ADACEL™ Vaccine Group 1: Adults 18 to 64 years of age received a single booster dose of Tdap vaccine (ADACEL™)
- ADACEL™ Vaccine Group 2: Children 4 to 8 years of age received a single booster dose of Tdap vaccine (ADACEL™)
- Total: Total of all reporting groups
Arm/Group | ADACEL™ Vaccine Group 1 | ADACEL™ Vaccine Group 2 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 20 | 20
  Between 18 and 65 years | 20 | 0 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (14.4) | 5.8 (1.1) | 25.0 (21.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 10 | 6 | 16
Region of Enrollment [Number; unit: Participants]
  China | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Adverse Events and Grade 3 Adverse Reactions Following a Single Booster Dose of Adacel™ Vaccine
Description: Solicited injection site reactions: Pain, Erythema, and Swelling; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia.
  China Food and Drug Administration (CFDA)-defined Grade 3 solicited reactions: Pain, incapacitating, unable to perform usual activities (Children, Group 2) and significant, prevents daily activity (Adults, Group 1); All Participants, Erythema and Swelling >30 mm; Fever (temperature) >39˚C; Headache, Malaise, and Myalgia, significant, prevents daily activity.
Time Frame: Day 0 up to Day 28 post-vaccination
Population: Serious adverse events and solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Groups:
- ADACEL™ Vaccine Group 1: Adults 18 through 64 years of age received a single booster dose of Tdap vaccine (ADACEL™)
- ADACEL™ Vaccine Group 2: Children 4 through 8 years of age received a single booster dose of Tdap vaccine (ADACEL™)
Arm/Group | ADACEL™ Vaccine Group 1 | ADACEL™ Vaccine Group 2
Number analyzed (Participants) | 20 | 20
Participants
  Grade 3 Injection site Pain | 0 | 0
  Grade 3 Injection site Erythema | 0 | 3
  Grade 3 Injection site Swelling | 0 | 3
  Grade 3 Fever | 0 | 0
  Grade 3 Headache | 0 | 0
  Grade 3 Malaise | 0 | 0
  Grade 3 Myalgia | 0 | 0
  Serious adverse events | 0 | 0

2. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reaction Following a Single Booster Dose of Adacel™ Vaccine
Description: as for outcome 1
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | ADACEL™ Vaccine Group 1 | ADACEL™ Vaccine Group 2
Number analyzed (Participants) | 20 | 20
Participants
  Injection site Pain | 6 | 9
  Grade 3 Injection site Pain | 0 | 0
  Injection site Erythema | 1 | 9
  Grade 3 Injection site Erythema | 0 | 3
  Injection site Swelling | 3 | 9
  Grade 3 Injection site Swelling | 0 | 3
  Fever | 0 | 3
  Grade 3 Fever | 0 | 0
  Headache | 1 | 1
  Grade 3 Headache | 0 | 0
  Malaise | 0 | 0
  Grade 3 Malaise | 0 | 0
  Myalgia | 1 | 1
  Grade 3 Myalgia | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination.
Arm/Group | ADACEL™ Vaccine Group 1 | ADACEL™ Vaccine Group 2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 9/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADACEL™ Vaccine Group 1 (N=20) | ADACEL™ Vaccine Group 2 (N=20)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Injection site Pain (General disorders) | 6 (6) | 9 (9)
Injection site Erythema (General disorders) | 1 (1) | 9 (9)
Injection site Swelling (General disorders) | 3 (3) | 9 (9)
Fever (General disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications